CLINICAL TRIAL: NCT07371520
Title: Application of Quantitative Hemorrhage Detection in Fetomaternal Hemorrhage Syndrome for the Diagnosis of Hemolytic Disease of the Newborn
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: IIT2025-275
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Hemolytic Disease of the Newborn
MeSH Terms: conditions — Erythroblastosis, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (2):
- Fetomaternal hemorrhage (FMH) values ≥ 0.5%
- Fetomaternal hemorrhage (FMH) value < 0.5%

SUMMARY:
This study adopted a single-center, prospective, observational study design. A consecutive cohort of pregnant and postpartum women who met the inclusion criteria was recruited from Shanghai First People's Hospital between January 2026 and December 2028. Quantitative hemorrhage detection was performed using residual clinical blood samples, and the diagnostic value of this detection for hemolytic disease of the newborn (HDN) was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age: Singleton pregnant women with gestational age ≥ 20 weeks.
* Clinical High-Risk Factors (meeting at least one of the following criteria):
* Traumatic Factors: Abdominal trauma (e.g., traffic accident, fall), intrauterine fetal version, amniocentesis, chorionic villus sampling (CVS).
* Obstetric Complications: Placental abruption, placenta previa, preeclampsia, unexplained antenatal hemorrhage, post-interventional therapy for twin-twin transfusion syndrome (TTTS).
* Fetal Abnormalities: Fetal growth restriction (FGR), unexplained abnormal fetal heart rate monitoring, fetal hydrops, fetal anemia (elevated middle cerebral artery peak systolic velocity (MCA-PSV) detected by Doppler ultrasound).
* High-Risk Population with Maternal-Fetal Blood Group Incompatibility: Maternal-fetal ABO or Rh-negative blood group incompatibility; positive result of the first-trimester antenatal antibody screening in pregnant women.

Exclusion Criteria:

* Pregnant women complicated with severe hematological diseases (e.g., coagulation disorders, immune thrombocytopenic purpura) or autoimmune diseases.
* Newborns who withdrew treatment for non-study-related reasons or were lost to follow-up after birth, resulting in missing outcome data.
* Termination of pregnancy due to various causes.
* Failure to complete the analysis due to unqualified core clinical data (e.g., quantitative hemorrhage test results, bilirubin levels) or unsatisfactory specimens (hemolysis, insufficient volume).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Pregnant and postpartum women
  2. Newborn
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemolytic Disease of the Newborn（HDN） | within 72 hours after birth
  All the following criteria must have been met for a diagnosis of HDN: (1) Blood group incompatibility between the mother and newborn; (2) hyperbilirubinemia with a positive direct antiglobulin test (DAT) result or hyperbilirubinemia with a negative DAT result and a positive elution testing result with high suspicion of a hemolytic condition such as anemia and/or reticulocytosis.

SECONDARY OUTCOMES:
Anemia: hemoglobin | within 72 hours after birth
  Hemoglobin Concentration in Peripheral Blood of Neonates
Incidence of severe hyperbilirubinemia | 30 days
  The peak concentration of serum bilirubin is more than the exchange criteria of same gestational age and day age group

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No